CLINICAL TRIAL: NCT02948010
Title: CPAP Device In-lab Assessment NZ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CIA187
Record Dates: First submitted 2016-10-26; First posted 2016-10-28 (Estimated); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (9):
- Auto CPAP + comfort feature A (Active Comparator): Auto CPAP with comfort feature A using Fisher & Paykel Healthcare CPAP Device
  Interventions: Device: Auto CPAP + comfort feature A
- Auto CPAP with comfort feature B (Active Comparator): Auto CPAP with comfort feature B using Fisher & Paykel Healthcare CPAP Device
  Interventions: Device: Auto CPAP with comfort feature B
- Auto CPAP with no comfort feature (Active Comparator): Auto CPAP with no comfort feature using Fisher & Paykel Healthcare CPAP Device
  Interventions: Device: Auto CPAP with no comfort feature
- Auto CPAP with comfort feature A+B (Active Comparator): Auto CPAP with comfort feature A+B using Fisher & Paykel Healthcare CPAP Device
  Interventions: Device: Auto CPAP with comfort feature A+B
- CPAP with comfort feature A (Active Comparator): CPAP with comfort feature A using Fisher & Paykel Healthcare CPAP Device
  Interventions: Device: CPAP with comfort feature A
- CPAP with comfort feature B (Active Comparator): CPAP with comfort feature B using Fisher & Paykel Healthcare CPAP Device
  Interventions: Device: CPAP with comfort feature B
- CPAP with no comfort feature (Active Comparator): CPAP with no comfort feature using Fisher & Paykel Healthcare CPAP Device
  Interventions: Device: CPAP with no comfort feature
- CPAP with comfort feature A + B (Active Comparator): CPAP with comfort feature A + B using Fisher & Paykel Healthcare CPAP Device
  Interventions: Device: CPAP with comfort feature A + B
- CPAP at Sub therapeutic level (Active Comparator): CPAP at Sub therapeutic level using Fisher & Paykel Healthcare CPAP Device
  Interventions: Device: CPAP at Sub therapeutic level

INTERVENTIONS:
Device: Auto CPAP + comfort feature A — Auto CPAP + comfort feature A using Fisher & Paykel Healthcare CPAP Device
  Arms: Auto CPAP + comfort feature A
Device: Auto CPAP with comfort feature B — Auto CPAP with comfort feature B using Fisher & Paykel Healthcare CPAP Device
  Arms: Auto CPAP with comfort feature B
Device: Auto CPAP with no comfort feature — Auto CPAP with no comfort feature using Fisher & Paykel Healthcare CPAP Device
  Arms: Auto CPAP with no comfort feature
Device: Auto CPAP with comfort feature A+B — Auto CPAP with comfort feature A+B using Fisher & Paykel Healthcare CPAP Device
  Arms: Auto CPAP with comfort feature A+B
Device: CPAP with comfort feature A — CPAP with comfort feature A using Fisher & Paykel Healthcare CPAP Device
  Arms: CPAP with comfort feature A
Device: CPAP with comfort feature B — CPAP with comfort feature B using Fisher & Paykel Healthcare CPAP Device
  Arms: CPAP with comfort feature B
Device: CPAP with no comfort feature — CPAP with no comfort feature using Fisher & Paykel Healthcare CPAP Device
  Arms: CPAP with no comfort feature
Device: CPAP with comfort feature A + B — CPAP with comfort feature A + B using Fisher & Paykel Healthcare CPAP Device
  Arms: CPAP with comfort feature A + B
Device: CPAP at Sub therapeutic level — CPAP at Sub therapeutic level using Fisher & Paykel Healthcare CPAP Device
  Arms: CPAP at Sub therapeutic level

SUMMARY:
The purpose of this trial is to assess device performance against participants in an overnight study to ensure the product meets user and clinical requirements

DETAILED DESCRIPTION:
Existing Adult Continuous Positive Airway Pressure (CPAP) therapy users will be recruited for an overnight polysomnography (PSG) sleep study. The participants will use the investigational CPAP device and be connected to a PSG during their session. The device performance during the session will be assessed. Outcomes of the clinical investigation include downloadable device data reports, device error reports and participants perception questionnaires and PSG data.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Diagnosed with OSA by a practicing physician and prescribed PAP therapy (fixed or auto CPAP)
* Fluent in spoken and written English.

Exclusion Criteria:

* Be contraindicated for PAP (fixed or auto CPAP) therapy.
* Have another significant sleep disorder(s) (e.g. periodic leg movements or insomnia).
* Have obesity hypoventilation syndrome or congestive heart failure.
* Require supplemental oxygen with your PAP (fixed or auto CPAP) device.
* Have any implanted electronic medical devices (e.g. cardiac pacemakers).
* Be pregnant or think they might be pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2016-11; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Apnea Hypopnea Index (AHI) (i.e. number of events/hour). | 4 months
  Obtained from device and PSG data
Log of safety-related events, measured as number of safety-related faults | 4 months
  Obtained from device
Machine reported faults, measured as number of machine faults | 4 months
  Obtained from device

SECONDARY OUTCOMES:
Participant perception of the device, as determined by the questionnaire responses | 4 months
  Obtained through user questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Fisher & Paykel Healthcare, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No